CLINICAL TRIAL: NCT00273260
Title: The Effect on Behavior and Bone Mineral Density of Individualized Bone Mineral Density Feedback and Educational Interventions in Premenopausal Women: a Randomized Controlled Trial.
Brief Title: The Effectiveness of Individualised Bone Density Feedback and Osteoporosis Education in Premenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menzies Institute for Medical Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MRI-001
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2006-05-09 (Estimated); Status verified 2006-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Educational Status

INTERVENTIONS:
Behavioral: individualised bone density feedback and education

SUMMARY:
The purpose of this study is to determine whether giving women feedback concerning their bone mineral density, combined with either an information leaflet or group education concerning osteoporosis changes women's behavior and/or bone density.

DETAILED DESCRIPTION:
Fractures due to osteoporosis are a major public health problem. Bone density is one of the major predictors of these osteoporotic fractures and is the result of the amount of bone gained in early life (i.e peak bone mass) and subsequent bone loss. Cigarette smoking, physical inactivity and inadequate calcium intake are widely regarded as risk factors for osteoporosis (as well as for other common diseases for the former two). Despite this information being widely available and actively promoted, the prevalence of these risk factors in the population remains unacceptably high. In women (mean age 33) taking part in a study of the determinants of bone mass in children, we recently reported substantial change in these behaviours at 12 months follow-up when women received an information leaflet and individualised bone density feedback. These women were highly selected and it is unclear if this response is representative of all women. With this study, we aim to test whether individualised bone density feedback, combined with either an information leaflet or small group education will change women's osteporosis preventive behaviors and/or bone density.

Specifically, we aimed to test the following hypotheses:

1. Women are more likely to change calcium intake and physical activity if their BMD is low.
2. Group education (in the form of the Osteoporosis Prevention and Self Management course) will be more efficacious at changing these lifestyle behaviours than an information leaflet alone.
3. Bone density feedback and educational intervention have independent effects on behavior and BMD change.
4. Women who improve their physical activity or dietary calcium intake will have a change in bone mass over 2 years that is 0.34-0.54% per annum better (depending on site and lifestyle factor) than those who do not alter their behaviour.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 25 and 44 years of age

Exclusion Criteria:

* previous had measurement of bone densitometry
* thyroid disease
* renal failure
* malignancy
* rheumatoid arthritis
* history of hysterectomy
* hormone replacement therapy
* were pregnant or planning pregnancy within 2 years of study entry
* lactating.

Ages: 25 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400
Dates: Start 2000-01; Study Completion 2002-12

PRIMARY OUTCOMES:
Bone mineral density

SECONDARY OUTCOMES:
physical activity
dietary calcium intake
calcium supplement use
smoking status

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Jones, MD, Principal Investigator — Menzies Institute for Medical Research
Locations (1):
- Menzies Research Institute, Hobart, Tasmania, Australia

REFERENCES:
- [Background] Winzenberg TM, Oldenburg B, Frendin S, De Wit L, Jones G. A mother-based intervention trial for osteoporosis prevention in children. Prev Med. 2006 Jan;42(1):21-6. doi: 10.1016/j.ypmed.2005.11.006. Epub 2005 Dec 5. PMID 16336993
- [Result] Winzenberg TM, Oldenburg B, Frendin S, De Wit L, Jones G. Effects of bone density feedback and group education on osteoporosis knowledge and osteoporosis self-efficacy in premenopausal women: a randomized controlled trial. J Clin Densitom. 2005 Spring;8(1):95-103. doi: 10.1385/jcd:8:1:095. PMID 15722593
- [Result] Winzenberg TM, Riley M, Frendin S, Oldenburg B, Jones G. Sociodemographic factors associated with calcium intake in premenopausal women: a cross-sectional study. Eur J Clin Nutr. 2005 Mar;59(3):463-6. doi: 10.1038/sj.ejcn.1602105. PMID 15674306
- [Result] Winzenberg TM, Oldenburg B, Frendin S, Jones G. The design of a valid and reliable questionnaire to measure osteoporosis knowledge in women: the Osteoporosis Knowledge Assessment Tool (OKAT). BMC Musculoskelet Disord. 2003 Jul 24;4:17. doi: 10.1186/1471-2474-4-17. PMID 12877751
- [Result] Winzenberg T, Oldenburg B, Frendin S, De Wit L, Riley M, Jones G. The effect on behavior and bone mineral density of individualized bone mineral density feedback and educational interventions in premenopausal women: a randomized controlled trial [NCT00273260]. BMC Public Health. 2006 Jan 23;6:12. doi: 10.1186/1471-2458-6-12. PMID 16430773
- [Derived] Wu F, Wills K, Laslett LL, Riley MD, Oldenburg B, Jones G, Winzenberg T. Individualized Fracture Risk Feedback and Long-term Benefits After 10 Years. Am J Prev Med. 2018 Feb;54(2):266-274. doi: 10.1016/j.amepre.2017.10.018. Epub 2017 Dec 13. PMID 29246678
- [Derived] Wu F, Wills K, Laslett LL, Oldenburg B, Seibel MJ, Jones G, Winzenberg T. Cut-points for associations between vitamin D status and multiple musculoskeletal outcomes in middle-aged women. Osteoporos Int. 2017 Feb;28(2):505-515. doi: 10.1007/s00198-016-3754-9. Epub 2016 Sep 9. PMID 27631092
- [Derived] Wu F, Callisaya M, Laslett LL, Wills K, Zhou Y, Jones G, Winzenberg T. Lower limb muscle strength is associated with poor balance in middle-aged women: linear and nonlinear analyses. Osteoporos Int. 2016 Jul;27(7):2241-2248. doi: 10.1007/s00198-016-3545-3. Epub 2016 Feb 26. PMID 26919994